CLINICAL TRIAL: NCT07346924
Title: Probiotics as a Promising Adjunct: Improving Fatigue, Quality of Life, Disability, Mood and Inflammatory Markers in Relapsing-Remitting Multiple Sclerosis: A Randomized, Double-blind, Controlled Study
Brief Title: Effect of Probiotics on Relapsing-Remitting Multiple Sclerosis
Acronym: PRO-RRMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Foraysa Mohammed Talaat, Faculty of medicine, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-221-2023
Record Dates: First submitted 2025-12-25; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis (MS) Relapsing Remitting
Keywords: fatigue; depression; disability
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Fatigue; Depression | interventions — Yogurt

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Active Comparator): probiotic dietary supplements
  Interventions: Dietary Supplement: Probiotic dietary supplement
- Controlled group (Placebo Comparator): standard treatment only
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Dietary Supplement: Probiotic dietary supplement — The probiotic group only had regular daily probiotic intake in the form of 2 cups of yogurt rich in probiotics - each cup 105 gram containing 5 to 10 billion Colony forming unit (CFU)/mg of Bifidobacterium animalis DN-173 010, Bifidobacterium lactis DN 173 010, Bifidobacterium lactis CNCM 1-2494, Lactobacillus bulgaricus, Streptococcus thermophiles, Lactococcus lactis and yeast tablets 400 mg one tablet per day for each patient each tablet containing 6 billion CFU/mg of probiotics Saccharomyces cerevisiae and Saccharomyces boulardii, along 3 months from the start of the study
  Other Names: yogurt
  Arms: Probiotic Group
Other: Standard medical treatment — standard medical treatment
  Arms: Controlled group

SUMMARY:
This study aimed to assess the effect of probiotic supplementation on fatigue, quality of life, disability, depression and inflammatory markers in patients with relapsing-remitting multiple sclerosis (RRMS).

Patients were randomized to receive probiotics plus standard therapy The study sought to determine whether modulation of gut microbiota could provide additional clinical and immunological benefits in RRMS management.

DETAILED DESCRIPTION:
This trial was conducted as part of a Doctoral (PhD) thesis at the Department of Neurology, Cairo University

The purpose of the trial was to evaluate the potential effects of probiotic supplementation on clinical and biological outcomes in patients with relapsing-remitting multiple sclerosis (RRMS).

Multiple sclerosis is a chronic inflammatory and demyelinating disease of the central nervous system, in which immune dysregulation and gut microbiota imbalance may play a key role.

Recent evidence suggests that probiotics could exert beneficial immunomodulatory and anti-inflammatory effects, potentially improving patient outcomes.

In this randomized controlled study, patients with RRMS received either probiotic supplementation or standard therapy alone for a defined period.

The primary outcomes included changes in fatigue quality of life, disability and depressive symptoms Secondary outcomes included alterations in inflammatory biomarkers such as cytokines and other immune mediators.

The results of this study are expected to provide additional insights into the role of gut microbiota modulation as an adjunctive approach in the management of multiple sclerosis.

No major protocol deviations occurred, and the study adhered to ethical standards approved by the local ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite MS patients with a diagnosis of relapsing remitting multiple sclerosis according to revised McDonald criteria 2017.
* EDSS score of ≤ 4

Exclusion Criteria:

* Progressive MS either; primary progressive MS or secondary progressive MS
* Patients who had relapses and glucocorticoid therapy within the past 30 days.
* Pregnancy and women who were lactating within the prior six month
* Patients taking antibiotics
* History of gastroenteritis and bowel surgery over the past month, inflammatory bowel disease
* Presence of diabetes (type I & type II) or diseases causing significant nutritional status impairment (malignancy, chronic infections)
* Patients who have changed their disease modifying drugs in the past 6 months prior to study
* Impaired cognition that limited ability to complete the questionnaires. Addiction to drugs or alcohol.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with improving in fatigue | 3 months
  changes in fatigue status using modified fatigue impact scale which range from 0 to 84 where high scores worse outcome

SECONDARY OUTCOMES:
Inflammatory biomarkers | 3 months
  alterations in inflammatory biomarkers such as cytokines and other immune mediators

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No